CLINICAL TRIAL: NCT05742100
Title: Use of Darvadstrocel (Allogenic Stem Cell Therapy) for Crohn's Fistula in Real Clinical Practice: the National Project to Implement Mesenchymal Stem Cell for the Treatment of Perianal Crohn's Fistula (the PRIME Study)
Brief Title: Darvadstrocel for Crohn's Fistula in the Realworld
Status: Completed | Type: Observational
Sponsor: Dolores Herreros Marcos (Other)
Responsible Party: Sponsor-Investigator, Dolores Herreros Marcos, Principal Investigator, Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Organization: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Other Study IDs: Darvastrocel Prime Study 001
Record Dates: First submitted 2023-02-10; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Crohn's Fistula
Keywords: Adipose-derived stem cells; Cell therapy; Compassionate use; Crohn's disease; Fistula-in-ano
MeSH Terms: conditions — Crohn Disease; Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group of patients treated with darvadstrocel
  Interventions: Drug: Darvadstrocel

INTERVENTIONS:
Drug: Darvadstrocel — expanded allogeneic adipose-derived mesenchymal stem cell therapy for the treatment of complex perianal fistulas

SUMMARY:
Background Perianal fistula may affect 15-50% of patients with Crohn's disease (CD). Treatment is complex, requiring a multidisciplinary approach. Darvadstrocel (allogeneic mesenchymal cells obtained from lipoaspirates) was approved in 2018 by the European Medicines Agency and Spanish Agency of Medicines and Medical Products as a treatment for fistulas in CD. Recent European Crohn's and Colitis Organisation (ECCO) andSpanish Working Group on Crohn's Disease and Ulcerative Colitis (GETECCU) guidelines state that darvadstrocel is effective with a favourable safety profile,with a strong level of evidence (level 2).With this study we want to see the real efficacy of darvadstrocel in a Spanish population after 6 months of follow-up.

DETAILED DESCRIPTION:
Methods: The criteria for the Spanish National Health System to fund darvadstrocel treatment are: 1)complex fistula in a patient with CD; 2)failure of conventional and anti-tumour necrosis factor treatment; and 3)absence of collection s>2cm confirmed by pelvic MRI scan at the time of surgery. From November 2019 to April 2022, 73 patients were treated with darvadstrocel at 14Spanish centres and evaluated clinically and radiologically 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1)complex fistula in a patient with CD
* 2)failure of conventional and anti-tumour necrosis factor treatment
* 3)absence of collection s>2cm confirmed by pelvic MRI scan at the time of surgery

Exclusion Criteria:

* Patients with a diagnosis of rectovaginal fistula, rectal stenosis or severe active proctitis were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with complex anorectal fistulas associated with CD treated with darvadstrocel in the 14 dedicated centres from 29 November 2019 to 21 April2022 will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants with clinical remission | 6-month
  Clinical remission was defined as closure of all previously draining external openings treated with darvadstrocel, despite gentle finger compression
Number of Participants with clinical response | 6-month
  Clinical response was defined as closure of ≥50% of previously draining external openings treated with darvadstrocel, despite gentle finger compression
Number of Participants with clinical radiographic healing | 6-month
  Complete radiographic healing was defined as an MRI result with no fluid collection >2cm in all dimensions, no oedema and no inflammation nor sign of active inflammatory response;a remnant fistula tract scar may remain
Number of Participants with combined clinical-radiological response | 6-month
  Combined clinical-radiological response, a new concept, was used to describe patients who achieved both clinical remission and complete radiological healing.

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Herreros, Principal Investigator — Hospital Fundación Jiménez Diaz
Locations (1):
- Fundacion Jimenez Diaz, Madrid, Spain

REFERENCES:
- [Derived] Herreros MD, Ramirez JM, Otero-Pineiro AM, Marti-Gallostra M, Badiola I, Enriquez-Navascues JM, Millan M, Barreiro EM, De La Portilla F, Suarez Alecha J, Garcia-Olmo D; National Project to Implement Mesenchymal Stem Cell for the Treatment of Perianal Crohn's Fistula (the PRIME Study) Group. Use of Darvadstrocel (Allogenic Stem Cell Therapy) for Crohn's Fistulas in Real Clinical Practice: The National Project to Implement Mesenchymal Stem Cell for the Treatment of Perianal Crohn's Fistula (the PRIME Study). Dis Colon Rectum. 2024 Jul 1;67(7):960-967. doi: 10.1097/DCR.0000000000003216. Epub 2024 Apr 11. PMID 38603800